CLINICAL TRIAL: NCT06539273
Title: Effectiveness of Exosome Treatment in Androgenetic Alopecia - Outcomes of a Prospective Study
Brief Title: Exosome Treatment in Androgenetic Alopecia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yeditepe University Hospital (Other)
Responsible Party: Principal Investigator, Mert Ersan, Asst.Prof., Yeditepe University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YeditepeKAEK1809
Record Dates: First submitted 2024-08-01; First posted 2024-08-06 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Androgenetic Alopecia; Exosomes
Keywords: androgenetic alopecia; exosome; extracellular vesicles; hair density; hair loss; mesenchymal stromal cells
MeSH Terms: conditions — Alopecia | interventions — Exosome Multienzyme Ribonuclease Complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): Intervention group
  Interventions: Drug: Exosome Complex, RNA

INTERVENTIONS:
Drug: Exosome Complex, RNA — A total of 3 mL of exosomes (2 mL to the frontal and 1 mL to the vertex region) was injected using napage technique (10¹⁰ extracellular vesicles in 1 mL)

SUMMARY:
This study aims to elucidate the effect of "foreskin-derived mesenchymal stromal cells derived exosome" injection into the scalp on hair density in patients with androgenetic alopecia and the contribution of this treatment on patient satisfaction.

DETAILED DESCRIPTION:
Within the scope of this research, we aim to elucidate the effect of "foreskin-derived mesenchymal stromal cells derived exosome" injection into the scalp on hair density in patients with androgenetic alopecia and the contribution of this treatment on patient satisfaction.This prospective study included 30 male patients, aged between 22 and 65, with hair type III-VI according to the Norwood-Hamilton scale, who agreed not to change their hairstyle and would not undergo any hair care or treatment during the study.Foreskin-derived Mesenchymal Stem Cells (MSCs) were utilized, sourced from the Extracellular Vesicle and Exosome Research Laboratory (EVER Lab) at Yeditepe University.The cell culture media is collected from a combination of FBS and antibiotic-free stem cell culture. An ATPS-Exosome isolation solution is prepared by blending Polyethylene glycol (PEG) and Dextran (DEX) at a 7.7:3.3 (w/w) ratio with distilled water.

Stem cell exosome concentration measurement and determination of exosome size and density distribution were conducted using Nanosight NS300 (Malvern Instruments) equipped with a 488 nm laser.Exosomal surface antigens were assessed using Flow Cytometry.

Before the exosome injections of 30 male patients with androgenetic alopecia, frontal and vertex regions where hair loss occurred on the scalp were imaged with a digital camera.An area of 1 cm2 from each of the mentioned areas were selected and 40x magnification images of those areas were taken with digital dermatoscopyUsing these dermatoscopic images, hair densities (hair count/cm2) were recorded with Trichoscan (TrichoLab GmbH, Germany). The patients were called for control at the 4th and 12th weeks after the injection. During these sessions, photographs of the same areas were taken with the same digital camera, from the same distance and under the same light and flash (1/200 s; f/6,3; ISO 160). During the controls, same topographic points were found (2 frontal and 1 vertex points) and these areas were imaged with digital dermatoscopy under x40 magnification. Hair densities were recorded with Trichoscan analyses and the averages of the 3 treated areas were taken.

Additionally, at the 4- and 12-week check-ups, a hair growth survey, as defined by Barber at al, was modified and administered to the patients [8]. In this modified survey, patients were asked 2 questions. Question one was "Has your hair loss decreased?" while the second question was "Have you noticed new hair growing?"

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged between 22 and 65, with hair type III-VI according to the Norwood-Hamilton scale,
* Patients who agreed not to change their hairstyle and would not undergo any hair care or treatment during the study

Exclusion Criteria:

* Patients using finasteride, dutasteride, steroids, vasodilators, anticonvulsants, beta-receptor blockers, bronchodilators, diuretics, spironolactone, cimetidine, diazoxide, cyclosporine, ketoconazole
* Patients with a history of surgery for hair loss, such as hair transplantation or scalp reduction
* Patients with a history of topical steroids or hair growth solutions for hair within the last year
* Patients with uncontrolled blood pressure and blood sugar levels in the last 6 months, infectious skin diseases or psychiatric disorders, a history of treatment of hyperthyroidism or hypothyroidism, aspartate aminotransferase (AST) or alanine aminotransferase (ALT) serum levels >80 mg/dL or creatinine (Cr) level >1.5 mg/dL
* Patients who were actively pregnant, breastfeeding, or planning to become pregnant within the next 6 months

Ages: 22 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients with androgenetic alopecia
Enrollment: 30 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-05 (Actual)

PRIMARY OUTCOMES:
Hair density | 4th and 12th weeks
  Increase in hair density (number of hair/cm2)

SECONDARY OUTCOMES:
Patient satisfaction survey | 4th and 12th weeks
  Increase Patient satisfaction in 4th and 12th weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Yeditepe University Kozyatagi Hospital, Istanbul, Atasehir, Turkey (Türkiye)